CLINICAL TRIAL: NCT01502579
Title: An Observational Study of the Relationship Between Pathological Variants and Clinical Data at Presentation and Follow-up in IgA Nephropathy
Brief Title: An Observational Study of IgA Nephropathy: Pathological Variants and Clinical Data
Status: Completed | Type: Observational
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Wei Shi, Professor, Guangdong Provincial People's Hospital
Other Study IDs: GGH201106
Record Dates: First submitted 2011-12-29; First posted 2011-12-30 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: IgA Nephropathy
Keywords: IgA nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The pathological variants of IgA nephropathy identified by the Oxford classification may be related to the clinical data at presentation and follow-up, including proteinuria and renal function. This study is aimed to identify the potential relationship between pathological variants and clinical data in IgA nephropathy.

ELIGIBILITY:
Inclusion Criteria:

* biopsy-proven IgA nephropathy;

Exclusion Criteria:

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population from which the cohort will be selected is these who have received renal biopsy in Guangdong General Hospital
Sampling Method: Probability Sample
Enrollment: 603 (Actual)
Dates: Start 2011-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
glomerular filtration rate decline or end-stage renal disease or doubling of serum creatinine | after the biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Wei Shi, MD,PhD, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China